CLINICAL TRIAL: NCT00053625
Title: Deep Brain Stimulation for Parkinson's Disease Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS037959 (NIH)
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; deep brain stimulation; DBS
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SA #1 Arm 1: Unilateral DBS in GPi (Active Comparator)
  Interventions: Procedure: deep brain stimulation
- SA #1 Arm 2: Unilateral DBS in STN (Active Comparator)
  Interventions: Procedure: deep brain stimulation
- SA #2 Arm 1: Bilateral DBS in GPi (Active Comparator): Patients with GPi bilateral DBS (previously had unilateral DBS in the GPi, now have bilateral DBS in GPi)
  Interventions: Procedure: deep brain stimulation
- SA #2 Arm 2: Bilateral DBS in STN (Active Comparator): Patients with STN bilateral DBS (previously had unilateral DBS in the STN, now have bilateral DBS in STN)
  Interventions: Procedure: deep brain stimulation

INTERVENTIONS:
Procedure: deep brain stimulation — Deep brain stimulation (DBS) is a surgical intervention used to treat movement disorders such as Parkinson's disease (PD). Target sites of stimulation may differ among patients. The Gpi and STN are two commonly targeted sites within the brain for treatment of PD, yet differences in outcomes between stimulation at the Gpi vs the STN (unilateral and bilateral) are not currently well understood.
  Other Names: DBS

SUMMARY:
The purpose of this trial is to evaluate the effect of deep brain stimulation in the the globus pallidus (Gpi) and the subthalamic nucleus (STN) on motor, neuropsychological and psychiatric function, and quality of life in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Medical therapy is the mainstay of treatment for patients with Parkinson's disease (PD). After several years of drug therapy, however, a large proportion of patients experience worsening of their parkinsonism and develop incapacitating motor fluctuations and dyskinesias. To deal with this, attention has been directed to surgical procedures, such as deep brain stimulation (DBS). Recently, stimulating the areas of the brain that control movement, the globus pallidus (Gpi) and subthalamic nucleus (STN), has been proposed as a therapy for treating many of the disabling symptoms associated with PD and drug-induced side effects.

The major aim of this 5-year study is to carry out a prospective, double blinded, randomized, clinical trial of DBS for medically intractable PD. The study will evaluate the effect of DBS in the Gpi and STN on motor, neuropsychological and psychiatric function, and quality of life in patients with PD. The study also will address two key issues: 1) whether there are differences between unilateral Gpi-DBS and STN-DBS and 2) which patients are the best candidates for bilateral DBS.

ELIGIBILITY:
INCLUSION:

* Clinical diagnosis of Idiopathic Parkinson's Disease based on the presence of at least 2 of the cardinal motor signs (akinesia/bradykinesia, rigidity, tremor, and gait/balance disorder) and a clear response to levodopa therapy.
* Hoeh & Yahr staging III or worse "off " medication periods.
* Intractable, disabling motor fluctuations, dyskinesias, or freezing episodes.
* Unsatisfactory clinical response to maximal medical management or previous surgical treatment.
* Stable on Parkinson's medications for at least 30 days with total L-dopa equivalence varying no more than +/- twenty percent during the 30 day period.
* Absence of cognitive, or psychiatric or other co-morbidities that might interfere with the patient's ability to understand and sign the informed consent form.

EXCLUSION:

* Clinically significant medical history that increases pre- / post operative complications (Cardiac or pulmonary disease, uncontrolled hypertension, diabetes…).
* Secondary or atypical parkinsonism as suggested by: i. History of stroke, encephalitis, exposure to toxins or neuroleptics. ii. Neurologic signs of upper motor neuron or cerebella involvement, supranuclear gaze palsy, or significant autonomic dysfunction. iii. MRI scan with evidence of significant brain atrophy, lacunar infracts, or iron deposits in the putamen.
* Dementia as indicated by a Mattis Dementia Rating Scale (DRS) less than 116 or DSM-IV criterion for dementia.
* Clinically significant psychiatric disorder meeting Structured Clinical Interview for the DSM-IV criteria for an active anxiety, depressive, or psychotic disorder.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 1999-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean change in total UPDRS score (baseline to six-months post DBS surgery) | Followed for minimum of 5 years
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a commonly used survey tool used to assess symptom severity of patients with Parkinson's disease (PD). It covers several different domains including 1) thought, behavior and mood 2) activities of daily living 3) motor activity 4) complications of therapy and others. The mean change from baseline to six months after DBS surgery for patients with DBS in the GPi vs the STN will be compared after being adjusted for differences in age and time since PD diagnosis.

SECONDARY OUTCOMES:
Mean change in UPDRS subscales and individual scores | Baseline to 6 months
  Subscales include domains including behavior and mood, activities of daily living, motor function, complications of therapy and others.
  Individual scores to be evaluated include scores for tremor, rigidity, bradykensia, gait, and postural stability.
  Other secondary endpoints include: Hoehn and Yahr staging, Modified Schwab and England Scale, timed test results, scores from psychiatric and quality of life assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold L Vitek, M.D., Ph.D., Principal Investigator — Cleveland Clinic Foundation, Director - Functional Neuroscience Research Center; Mahlon R. DeLong, M.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University School of Medicine, Neurology Department, Atlanta, Georgia
  - Cleveland Clinic Foundation, Cleveland, Ohio